CLINICAL TRIAL: NCT00233220
Title: Multi-site Randomized Controlled Trial for Blood Pressure Control in Hypertensive African Americans
Brief Title: Blood Pressure Control in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Gbenga Ogedegbe, Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 322; R01HL078566 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients and doctors will take part in a multicomponent, multi-level intervention.
  Interventions: Behavioral: Multicomponent, multi-level intervention targeted at physicians and patients
- 2 (Active Comparator): Patients will receive usual care.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Multicomponent, multi-level intervention targeted at physicians and patients — The patient intervention will include an innovative patient education approach known as Self-Paced Programmed Instruction that will be used to educate patients on knowledge of HTN; behavioral counseling by trained C/MHC dieticians on lifestyle modification; and home BP monitoring to activate patients in their own care. The physician intervention comprises online continuing medical education (CME) courses on management of HTN based on the Joint National Committee-7 (JNC-7) guidelines; online HTN rounds or case conferences with HTN specialists; and feedback to physicians on clinical performance measures via computerized decision support systems. The intervention will be delivered to patients every 3 months during regular office visits for 12 months, while the physician intervention will occur every month for the duration of the trial.
  Arms: 1
Behavioral: Usual Care — Patients will receive usual care.
  Arms: 2

SUMMARY:
The purpose of this study is to test the effectiveness of a multi-component evidence-based intervention that targets both patients and physicians, in improving BP control rates in patients followed in 30 Community/Migrant Health Centers (C/MHCs).

DETAILED DESCRIPTION:
BACKGROUND:

African Americans (AA) have the highest prevalence of hypertension (HTN) in the U.S., with a resultant greater HTN-related mortality compared to whites. Barriers to BP Control in AA exist at 3 levels of care: the patient, the physician, and the healthcare system. Using the Chronic Care Model as a framework, the investigators seek to test the effect on BP control of a multicomponent, multi-level intervention targeted at physicians and patients.

DESIGN NARRATIVE:

Using the Chronic Care Model as a framework, the investigators seek to test the effect on BP control of a multicomponent, multi-level intervention targeted at physicians and patients. They will conduct a clustered randomized controlled trial in which 30 C/MHCs will be randomized to either the intervention or usual care. A total of 990 patients with uncontrolled HTN (BP greater than 140/90 mm Hg) will be enrolled for this trial. Components of the patient intervention include an innovative patient education approach known as Self-Paced Programmed Instruction that will be used to educate patients on knowledge of HTN; behavioral counseling by trained C/MHC dieticians on lifestyle modification; and home BP monitoring to activate patients in their own care. The physician intervention comprises online continuing medical education (CME) courses on management of HTN based on the Joint National Committee-7 (JNC-7) guidelines; online HTN rounds or case conferences with HTN specialists; and feedback to physicians on clinical performance measures via computerized decision support systems. The intervention will be delivered to patients every 3 months during regular office visits for 12 months, while the physician intervention will occur every month for the duration of the trial. Patients and physicians at the usual care C/MHCs will receive NHLBI patient education materials and print versions of JNC-7 guidelines respectively.

The primary outcome is the proportion of patients with adequate BP control at 12 months in each condition as defined by JNC-7 criteria (BP less than 130/80 mm Hg for patients with diabetes or kidney disease; and BP less than 140/90 mm Hg for all other patients). The secondary outcomes are within-patient change in systolic BP and diastolic BP from baseline to 12 months; the maintenance of the intervention effects one year after trial; and the cost effectiveness of the intervention at 12 months. The long-term goal of this project is to refine the intervention as a result of the data obtained and to develop a standardized protocol that can be integrated into the usual care procedures of the C/MHCs. Thus, maximizing the likelihood that the intervention will be translated into practice, at each of the participating Community Health Centers.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled Hypertension
* African American

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1039 (Actual)
Dates: Start 2004-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Control BP | Measured at Year 1

SECONDARY OUTCOMES:
Change in systolic BP and diastolic BP | Measured at Year 1
Maintenance of the intervention effects | Measured at Year 1
Cost effectiveness of the intervention | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Gbenga G Ogedegbe, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Ogedegbe G, Tobin JN, Fernandez S, Gerin W, Diaz-Gloster M, Cassells A, Khalida C, Pickering T, Schoenthaler A, Ravenell J. Counseling African Americans to Control Hypertension (CAATCH) trial: a multi-level intervention to improve blood pressure control in hypertensive blacks. Circ Cardiovasc Qual Outcomes. 2009 May;2(3):249-56. doi: 10.1161/CIRCOUTCOMES.109.849976. PMID 20031845
- [Background] Fernandez S, Tobin JN, Cassells A, Diaz-Gloster M, Kalida C, Ogedegbe G. The counseling African Americans to Control Hypertension (CAATCH) Trial: baseline demographic, clinical, psychosocial, and behavioral characteristics. Implement Sci. 2011 Sep 1;6:100. doi: 10.1186/1748-5908-6-100. PMID 21884616
- [Derived] Forsyth J, Schoenthaler A, Chaplin WF, Ogedegbe G, Ravenell J. Perceived discrimination and medication adherence in black hypertensive patients: the role of stress and depression. Psychosom Med. 2014 Apr;76(3):229-36. doi: 10.1097/PSY.0000000000000043. PMID 24677163
- [Derived] Ogedegbe G, Tobin JN, Fernandez S, Cassells A, Diaz-Gloster M, Khalida C, Pickering T, Schwartz JE. Counseling African Americans to Control Hypertension: cluster-randomized clinical trial main effects. Circulation. 2014 May 20;129(20):2044-51. doi: 10.1161/CIRCULATIONAHA.113.006650. Epub 2014 Mar 21. PMID 24657991